CLINICAL TRIAL: NCT01630252
Title: A Phase IIa Efficacy and Safety Study of PGL5001 Versus Placebo Administered for up to 5 Months With Concomitant Administration of Depot Medroxyprogesterone Acetate for the Treatment of Peritoneal and/or Ovarian Endometriosis With an Inflammatory Component.
Brief Title: PGL5001 Proof of Concept Study in Inflammatory Endometriosis
Acronym: JADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGL11-021
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — bentamapimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part A2 - Active Treatment arm (Active Comparator): PGL5001 for 8 weeks + one DMPA injection
  Interventions: Drug: PGL5001
- Part A2 - Placebo Treatment arm (Placebo Comparator): PGL5001 matching placebo for 8 weeks + one DMPA injection
  Interventions: Drug: Placebo
- Part B - Active treatment arm (Active Comparator): PGL5001 for 20 weeks + two DMPA injections
  Interventions: Drug: PGL5001
- Part B - Placebo Treatment arm (Placebo Comparator): PGL5001 matching placebo for 20 weeks + two DMPA 150mg injections
  Interventions: Drug: Placebo
- Part A1 - Active Treatment arm (Experimental): PGL5001 for 8 weeks + one unique DMPA 150 mg injection
  Interventions: Drug: PGL5001

INTERVENTIONS:
Drug: PGL5001 — PGL5001 320mg/day (160 mg twice a day) for 8 weeks + one unique DMPA 150 mg injection
  Arms: Part A2 - Active Treatment arm
Drug: Placebo — PGL5001 matching placebo (twice a day) for 8 weeks + one unique DMPA 150 mg injection
  Arms: Part A2 - Placebo Treatment arm
Drug: PGL5001 — PGL5001 320mg/day (160 mg twice a day) for 20 weeks + DMPA 150mg injection. Second DMPA injection between 85 to 89 days after first injection
  Arms: Part B - Active treatment arm
Drug: Placebo — PGL5001 matching placebo (twice a day) for 20 weeks + DMPA 150mg injection. Second DMPA injection between 85 to 89 days after first injection
  Arms: Part B - Placebo Treatment arm
Drug: PGL5001 — PGL5001 320mg/day (160 mg twice a day) for 8 weeks + one unique DMPA 150 mg injection
  Arms: Part A1 - Active Treatment arm

SUMMARY:
This is a prospective, three-part (Part A1, Part A2 and Part B),Phase II study investigating the efficacy, safety, pharmacokinetics and pharmacodynamics of the JNK inhibitor PGL5001 orally administered for up to 5 months with concomitant DMPA administration for the treatment of laparoscopically diagnosed inflammatory endometriosis. The part A1 is open-label, the parts A2 and B are double-blind.

The target population will be women of reproductive age and suffering from newly diagnosed peritoneal and/or ovarian endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* The Subject must provide written informed consent prior to initiation of any study related procedures.
* The Subject must be an adult woman of reproductive age, aged from 18 and above.
* The Subject must be a newly diagnosed patient suffering from peritoneal and/or ovarian endometriosis with at least 15% of the endometriotic lesions observed at the study diagnostic laparoscopy being red inflammatory lesions and with a proven histological diagnosis.
* The Subject must consent to the scheduling of a second laparoscopy for surgical treatment at the study end.
* The Subject must have a history of pelvic pain for at least 3 months prior to the screening visit.

Exclusion Criteria:

* The Subject is over 40 years old and has a FSH serum level during Day 2-4 of her cycle ≥ 21.5 mIU/ml.
* The Subject has a positive pregnancy test at baseline or is breast-feeding or planning a pregnancy during the course of the study.
* The Subject is known for having a cause of chronic abdominal/pelvic pain other than endometriosis (e.g. inflammatory bowel disease, fibromyalgia, interstitial cystitis).
* The Subject has a history of surgical treatment for endometriosis prior to the study diagnostic laparoscopy.
* The Subject is requiring urgent surgical excision of endometriotic lesions at the time of first diagnostic laparoscopy.
* The Subject has a history (in the past 12 months) of or a current medical treatment for endometriosis other than NSAID (e.g. GnRH agonist or antagonist, danazol, continuous oral combined oestroprogestogens).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of treatment in the number and percentage of red lesions (and/or inflammatory lesions), based on total number of red and black lesions. | at week 8, week 20

CONTACTS AND LOCATIONS:
Overall Officials: Elke Bestel, MD, Study Director — PregLem SA
Locations (1):
- Prywatna Klinika Połozniczo-Ginekologiczna Sp z o.o., Bialystok, Poland